CLINICAL TRIAL: NCT00284739
Title: Alteplase for Percutaneous Treatment of Loculated Abdominopelvic Abscesses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HI-03HYoon-02
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Results first posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Abdominal Abscess; Pelvic Abscess
MeSH Terms: conditions — Abdominal Abscess | interventions — Tissue Plasminogen Activator; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alteplase (Experimental): Multiple Alteplase injection into the abscess collection to improve percutaneous drainage
  Interventions: Drug: Alteplase
- Saline (Placebo Comparator): Multiple normal saline injection into the abscess collection to improve percutaneous drainage
  Interventions: Other: saline

INTERVENTIONS:
Drug: Alteplase — 2mg or 4mg given twice daily for three days into loculated abscess
  Other Names: Activase
  Arms: Alteplase
Other: saline — saline injection twice daily for three days
  Arms: Saline

SUMMARY:
Intracavitary injection of low dose alteplase into loculated abdominopelvic abscesses will reduce the duration of percutaneous drainage and increase the proportion of successful drainages.

DETAILED DESCRIPTION:
The use of fibrinolytics for the percutaneous drainage of loculated pleural effusions has been shown to reduce the catheter dwell time and to improve drainage of the effusions. Abscesses in the abdomen and pelvis are often loculated which makes percutaneous drainage difficult. We hypothesize that the infusion of alteplase via a drainage catheter into the loculated abscess collections of the abdomen and pelvis will similarly decrease catheter dwell time and improve overall abscess drainage. The direct injection of Activase into abscess cavities utilizes a very low dose of drug within a closed environment which should not be associated with any significant risk of hemorrhage. To date, there does not appear to be a significant risk of systemic hemorrhagic complications associated with the use of intracavitary thrombolytics for the drainage of abdominopelvic abscesses although only a few such studies have been reported. We hope to prove that the use alteplase for intracavitary thrombolysis improves outcomes associated with percutaneous catheter drainage of loculated abscess collections without increasing complications or costs.

The design of the trial will be as a single-center, prospective, open-label, randomized trial comparing the infusion of Activase versus saline for treatment of loculated abdominopelvic abscesses requiring percutaneous drainage. Patients with loculated abdominopelvic abscesses who are referred for percutaneous drainage will be eligible for this study. Patients will undergo standard placement of a 10-12 french percutaneous drain into their abscess cavity under computed tomography guidance. If the entire contents of the abscess cavity cannot be aspirated at the time of initial catheter placement, the abscess will be assumed to be loculated. The patient will then be randomized to have their abscess catheter irrigated twice a day with a volume of fluid approximately equal to the one-half the residual volume of the abscess. In the control group, the normal saline will be fluid instilled into the abscess cavity. The study group will receive Activase reconstituted in sterile water and then diluted to the appropriate volume with normal saline.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Age > 18 years
* Adult, non-gravid patients with loculated abdominopelvic abscesses immediately after percutaneous drainage will be eligible to participate. A loculated abscess is defined as an abscess whose contents cannot be completely drained at the time of initial catheter placement as documented on CT.

Exclusion Criteria:

* Active internal bleeding, involving intracranial and retroperitoneal sites, or the gastrointestinal, genitourinary, or respiratory tracts
* History of stroke within 6 months
* Uncorrectable bleeding diathesis (INR > 1.3 despite therapy)
* Recent intracranial or intraspinal surgery or trauma
* Pregnancy (positive pregnancy test)
* Pancreatic abscesses
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial
* Participation in another clinical investigation within previous 30 days of catheter placement
* Prior enrollment in the study
* Known allergy to Alteplase or any of its components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Chun Yoon, MD, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Foundation Hospital, Honolulu, Hawaii, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitalized patients with loculated abscess were enrolled
Pre-assignment Details: All patients had undergone percutaneous drainage for abscess and loculation documented by residual fluid surrounding the catheter after initial drainage
Period: Overall Study
Arm/Group | Alteplase | Saline
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alteplase | Saline | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 15
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (19) | 57 (20) | 52 (20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Requiring Surgical Debridement for a Persistent Abscess Within 30 Days Following Initial Drainage
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Alteplase | Saline
Number analyzed (Participants) | 11 | 9
participants | 3 | 7

2. Secondary Outcome: Percentage of Loculated Abscesses Which Completely Resolve With Percutaneous Drainage Alone at the First Follow-up CT Scan Performed 3 Days After Initial Drain Placement
Description: This is the percentage of participants in whom their loculated abscess completely resolve with percutaneous drainage at the time of the first followup CT performed at 3 days after start of the intervention and therefore do NOT require additional surgical intervention.
Time Frame: 3 days
Measure: Number; unit: percentage of patients
Arm/Group | Alteplase | Saline
Number analyzed (Participants) | 11 | 9
percentage of patients | 82 | 33

3. Secondary Outcome: Duration (in Days) of Percutaneous Drainage.
Description: The total number of days that the drainage catheter was left in place from the time of randomization until the time of catheter removal. The maximum duration of measurement for this outcome was up to 30 days.
Time Frame: Up to 30 days
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Alteplase | Saline
Number analyzed (Participants) | 11 | 9
days | 6 [4.5 to 7.5] | 11 [8 to 14]

ADVERSE EVENTS:
Arm/Group | Alteplase | Saline
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes